CLINICAL TRIAL: NCT00886548
Title: Echocardiographic Examination Performed by Nurses in Cardiac Intensive Care Unit. Is it Clinical Useful?
Brief Title: Echocardiographic Examination Performed by Nurses in Cardiac Intensive Care Unit
Status: Withdrawn | Type: Observational
Why Stopped: Delayed inclusion
Sponsor: Helse Nord-Trøndelag HF (Other)
Responsible Party: Sponsor
Other Study IDs: SL-20091
Record Dates: First submitted 2009-04-21; First posted 2009-04-23 (Estimated); Last update posted 2021-11-09 (Actual); Status verified 2021-11

CONDITIONS: Heart Failure; Myocardial Infarction; Pleural Effusion
MeSH Terms: conditions — Heart Failure; Myocardial Infarction; Pleural Effusion

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Ultrasound performed: Single arm study.
  Interventions: Procedure: Ultrasound performed

INTERVENTIONS:
Procedure: Ultrasound performed — Nurse-driven ultrasound performed

SUMMARY:
The purpose of this study is:

* To study the clinical usefulness of nurse-performed ultrasound and echocardiographic examinations in a cardiac intensive care unit.
* To study reproducibility of nurse-performed ultrasound and echocardiographic examinations in a cardiac intensive care unit.
* To study which ultrasound measure that best correlate with the amount of pleural effusion.

DETAILED DESCRIPTION:
For a period of 1 year patients in our cardiac intensive care unit will be recruited to nurse-drive ultrasound and echocardiographic examinations, after informed consent. Nurses underwent a training programme and their skills are approved by cardiologist. Our department does not always have a cardiologist on duty and indication for nurse-driven ultrasound examination is decided by the doctor responsible for the treatment, who not always are trained in echocardiography/ultrasound. We aim to study the described hypothesis.

ELIGIBILITY:
Inclusion Criteria:

* Patient at Cardiac intensive care unit, Levanger Hospital
* Doctor responsible for treatment finds echocardiographic/ultrasound examination indicated.

Exclusion Criteria:

* None

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients hospitalized at Cardiac Intensive Care Unit at Levanger Hospital
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2009-04; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Change of diagnosis | 6-12 months

SECONDARY OUTCOMES:
Change of treatment | 6-12 months
Quantification of pleural effusion | 6-12 months
Reproducibility of nurse-performed examinations | 6-12 months

CONTACTS AND LOCATIONS:
Overall Officials: Håvard Dalen, MD, Study Chair — Levanger Hospital, Nord-Trøndelag Health Trust
Locations (1):
- Department of Medicine, Hospital of Levanger, Levanger, Norway